CLINICAL TRIAL: NCT01825980
Title: Double-blind, Randomized, Placebo-controlled, Multi-center Trial to Determine the Safety and Antiviral Effect of 3 Days of BZF961 With or Without Ritonavir Boosting in Hepatitis C Virus (HCV) Infected Patients
Brief Title: Proof of Concept Study to Determine the Safety and Antiviral Effect of BZF961 With or Without Ritonavir Boosting in Hepatitis C Virus Infected Patients
Acronym: CBZF961X2201
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CBZF961X2201; 2012-003103-35 (EudraCT Number)
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — BZF961; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BZF961 (Experimental)
  Interventions: Drug: BZF961; Drug: Ritonavir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BZF961 — There will be 2 parts to the study: Part 1: BZF monotherapy. Part 2: Cohort IIa: BZF961 monotherapy at 3 TBD doses; Cohort IIb: BZF961 in combination with ritonavir at TBD doses.
  Arms: BZF961
Drug: Ritonavir — Ritonavir will be given as a boosting agent in Part 2, Cohort IIb in combination with BZF961
  Arms: BZF961
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the antiviral activity of 3 days of BZF961. To determine safety and tolerability of BZF961 in HCV patients. To evaluate pharmacokinetics of BZF961 in HCV patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed Male & female treatment naive subjects, age 18-60 years of age with Hepatitis C genotype-1. Subjects must weight at least 50kg to participate in the study, and must have a body mass index (BMI) within the range of 18-36 kg/m2 Able to communicate well with the investigator, to understand and comply with the study requirements.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer: or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.

Subjects that were previously treated for HCV infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HCV viral load | Day 3
  Viral load samples will be taken at Day 3.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 2 weeks
Total BZF961 concentration in plasma | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, San Antonio, Texas

REFERENCES:
- See also: Results for CBZF9612201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14326